CLINICAL TRIAL: NCT05316818
Title: The Efficacy and Toxicity of Triplet Regimen (FOLFOXIRI) Versus Doublet Regimen (FOLFOX or FOLFIRI) as First Line Treatment in Locally Advanced, Recurrent or Metastatic Colorectal Carcinoma.
Brief Title: Triplet (FOLFOXIRI) vs. Doublet (FOLFOX or FOLFIRI) Regimen as a 1st Line Treatment in Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Ahmed Khalil Hassan, Assistant lecturer of clinical oncology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-160317
Record Dates: First submitted 2022-03-07; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: First line chemotherapy; FOLFOXIRI; standard doublet; Efficacy; Toxicity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — FOLFOXIRI protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triplet regimen (FOLFOXIRI) (Experimental): The treatment planned consisted of irinotecan 160 mg/m² in 250 ml of NaCl 0.9% over 1 hr, followed by 85 mg/m² oxaliplatin in 250 ml dextrose 5% given concurrently with a 400 mg/m² leucovorin intra venous infusion in 250 ml dextrose 5% for 120 min, followed by 2400 mg/m² for 44-hr continuous infusion
  Interventions: Drug: FOLFOXIRI Protocol
- standard duplet regimen (FOLFOX or FOLFIRI) (Active Comparator): Regimen consisted of 180 mg/m² intravenous infusion of irinotecan for 60 min OR 85 mg/m² oxaliplatin day 1 only followed by a 200 mg/m² intra venous infusion of leucovorin for 120 min, a 400 mg/m² intravenous bolus of fluorouracil, and a 600 mg/m² continuous infusion of fluorouracil for 22 hr to be repeated on day 2
  Interventions: Drug: FOLFOXIRI Protocol

INTERVENTIONS:
Drug: FOLFOXIRI Protocol — Triplet chemotherapy regimen consists from active three cytotoxic agents aiming to improve outcomes

SUMMARY:
This is a prospective randomized phase II trial was done in clinical oncology department at Kasr Alainy hospital, Cairo university (NEMROCK) to evaluate the role of intensification of chemotherapy in the first line for treatment of metastatic colorectal carcinoma by adding third agent to standard doublet regimen on oncological outcomes & assess tolerance to the intensified treatment

DETAILED DESCRIPTION:
Patients with histologically proven adenocarcinoma of the colon or rectum, with unresectable measurable metastatic disease, were enrolled and randomized in a 1:1 ratio.

Patients were assigned to receive FOLFOXIRI (experimental arm) or FOLFIRI or FOLFOX4 (control arm) biweekly up to 12 cycles.

Randomization was done by enclosed envelope method Evaluation of the patients for surgical resection of residual metastases was done every 12 weeks. In the case of secondary resection of metastases, patients completed with the same chemotherapy regimen received before resection up to 12 cycles Maintenance therapy with capecitabine for 6 months was administered for patients who achieved complete or partial tumor response. In case of disease progression, second line chemotherapy was then administered in both groups until tumor progression, the occurrence of an unacceptable adverse event, or patient refusal

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven adenocarcinoma of the colon or rectum, with unresectable measurable metastatic disease
* No previous treatment for the metastatic disease was allowed, only previously fluoropyrimidine-based adjuvant chemotherapy was allowed if ended more than 6 months before enrollment in the study
* Adequate haematological parameters (leukocyte count of at least 3,500/mm₃, neutrophil count of at least 1,500/ mm and platelet count of at least 100,000/mm
* Adequate liver and renal function parameters (serum creatinine ≤ 1.3 mg/dL, serum bilirubin ≤ 1.5 mg/dL and AST, ALT and alkaline phosphatase 2.5 x upper normal values or less.
* Patient had no co-morbidity disease

Exclusion Criteria:

* Poor performance status 3-4 according to ECOG score, prior chemotherapy for advanced, recurrent or metastatic disease, other simultaneous malignancies and pregnant or lactating female

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months ( from staring treatment till finishing 12 cycles, each cycle every 2 weeks)
  the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria
Rate of adverse events | During the study treatment period till 30 days following the end of therapy
  Adverse events (haematological & non-haematological) were assessed before each cycle using the Common Terminology Criteria for Adverse Events version (CTCAE) 5.0, 2017 with scale from (G0-5) for each event.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 18 months
  the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. Documentation of disease progressive disease is defined as per RECIST 1.1 criteria based on investigator assessment
Overall survival time (OS) | 18 months
  Defined as the length of time from date of randomization to the date of death due to any cause or due to lost follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El AiniH, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No